CLINICAL TRIAL: NCT04628156
Title: An Observational Study Of Chronic Pain In a Greek Population of Children, Adolescents And Adults With Cerebral Palsy
Brief Title: Chronic Pain In a Greek Population With Cerebral Palsy
Acronym: CPPain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cerebral Palsy Greece - Open Door (Other)
Responsible Party: Sponsor
Other Study IDs: CPChronicPain
Record Dates: First submitted 2020-10-08; First posted 2020-11-13 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Cerebral Palsy
Keywords: Chronic Pain
MeSH Terms: conditions — Cerebral Palsy; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatients in Cerebral Palsy Greece - Open Door: Outpatients with a diagnosis of cerebral palsy

SUMMARY:
The aim of this observational, cross-sectional study is to effectuate a survey of chronic pain in a population of children, adolescents and adults with various forms of cerebral palsy in an educational and therapeutic setting in Athens, Greece. (Cerebral Palsy Greece-Open Door) Prevalence, intensity and localisation of pain will be associated to factors related to the functional and communicative limitations of the study's participants. The study also examines the agreement rate between different information sources and evaluation levels of chronic pain assessment in cerebral palsy (self-reports, caregiver questionnaires, observational check-lists administered by rehabilitation professionals, clinical evaluations by experts). A further research aim is to identify behavioural markers of chronic pain in individuals with cerebral palsy and a very limited communicative level.

DETAILED DESCRIPTION:
Increasing research evidence suggests that children, adolescents and adults with cerebral palsy belong to a population with a significantly high prevalence of chronic and recurrent pain that has a negative impact on their participation level and their quality of life.

Etiology of pain in CP covers a broad spectrum of reasons. First of all, individuals with CP might, like any other person, have problems with headache, periodic pain and other commonly encountered causes of pain. Pain emerging from muscles, joints and the skeleton are common. For some individuals increased muscle tone, spasticity or dystonia can be an important contributing factor for pain. This type of pain often referred to as musculoskeletal pain can be localized in the back, neck, foot/ankle, shoulder, knee, hip and arm. Gastro-intestinal pain often caused by gastro-oesophageal reflux secondary to changed muscular function in the oesophagus or lower oesophageal sphincter and spinal deformity (scoliosis) is another source to chronic pain. Furthermore many activities of daily living such as getting dressed, being lifted and daily assisted stretching can be painful. Finally dental pain caused by difficulties in maintaining good oral hygiene or gastro-oesophageal reflux (causing erosions to the dental enamel and secondary caries) needs special consideration (AACPDM Fact Sheet). Children with CP who are faced with chronic pain use fewer coping strategies and tend to rely on social support. In the case of individuals with cerebral palsy who do not have the ability to communicate because of disabilities caused by central or peripheral nervous system impairment, chronic and incidental acute pain can remain undetected and undertreated. Assessing pain in individuals with cerebral palsy encompasses particular methodological challenges. Pain assessment in individuals with cerebral palsy must take into account their verbal or non-verbal communication level. In that case by proxy (observational-behavioural) tools are necessary. In addition using observational tools to truly recognize pain expression one should also considered that a number of factors such as learned reaction to chronic pain are reported to influence more than others the display of the behavioural pain indicators included in certain tools of behavioural pain assessment.

The aim of our study is the screening and assessment of chronic pain in a population of children, adolescents and adults with various forms of cerebral palsy in a specific special needs educational and rehabilitation setting in Athens, Greece (Cerebral Palsy Greece- Open Door). Furthermore, the investigators will explore the possible connection of pain in cerebral palsy with factors such as severity of CP, age, gender, comorbidities developmental status and current health status. A significant percentage of the study population has limited communication abilities. Consequently, this cross-sectional observational study has to take into account the verbal and non-verbal communication level of the population's subjects when determining the most appropriate pain assessment procedure, differentiating between patients whose pain status will be assessed through self-report and patients whose pain status will be assessed through observational tools (check lists). In terms of their reliability both self-report and by proxy (observational) tools of pain assessment, share some evidence of strong agreement between them. The following procedures will be followed:

1. Assessment of the level of verbal and non verbal communication skills The ability of the subjects to give valid and reliable information concerning their pain status through meaningful verbal and non verbal communication will be evaluated according to their Communication Function Classification System -CFCS classification levels by trained speech therapists. Classification is based on the effectiveness of communication between a sender and receiver of information. CFCS considers the familiarity of individual communication partners. All ways of communicating are considered including speech, gesture, facial expression and augmentative and alternative communication. A person classified at Level I is a more able communicator than a person classified at Level V. According to CFCS classification 4 categories could be defined. These are A. Children with adequate communication B. Children with inadequate communication C. Adults with adequate communication and D. Adults with inadequate communication.
2. Classifications of the type cerebral palsy and functional level Type of cerebral palsy will be taken into account according to ICD codes (ICD-10 version 2016) and functional motor ability will be recorded using Gross Motor Function Classification System (GMFCS) and the Manual Ability Classification System (MACS). The GMFCS was used to assess the severity of a child's neuromotor impairment. Based on this instrument, children were grouped according to the following levels of severity: levels I and II refer to those children with lower functional impairment and that are able to walk without restrictions; level III refer to those children that need help; level IV/V includes the children that use assistive technology to ambulate. The GMFCS was assesses for its validity and reliability with satisfactory results. MACS describes how children with cerebral palsy (CP) use their hands to handle objects in daily activities. MACS includes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life. Level I includes children with minor limitations, while children with severe functional limitations will usually be found at levels IV and V.
3. Selection of the appropriate tools for the assessment of pain for each category Subjective reports of pain location and intensity through non verbal communication (pointing) from study participants will be collected using the Wong Baker FACES Pain Rating Scale (permission needed) and the Body Diagram screening tool. The Body Diagram was tested for content and concurrent validity and alternate forms reliability. This tool is rated as approaching well-established according to the evidence based psychometric properties assessment criteria. In terms of clinical utility this tool was classified as strong.

   Self-reports will be administered to subjects who have an adequate communication level (CFCS level I, II, III), following the directives set by relevant research. In the case of subjects with an adequate communication level (CFCS level I ,II, III) but an inadequate manual ability functional level (MACS level IV and V) the administration of Wong Baker FACES Pain Rating Scale and of the Human Form diagrams will be facilitated by the use of assistive technology.

   Pain observational reports by proxy (teacher, therapist in the rehabilitation setting) will be collected using translated versions of the Non Communicating Children's Pain Check List and the Non Communicating Adults' Pain Check List. These observational reports will be administered in the case of subjects with a CFCS level IV and V and a developmental age lower than 3 years old. The NCCPC-R (revised) version requires a 2-hour observational period followed by the completion of the 30-item questionnaire. The NCCPC-R hosts strong external validity as psychometric testing within natural and clinical settings. Researchers have affirmed the NCCPC-R accurately captures pain behaviours across various levels of a child's development.78 The working group recommended the NCCPC-R for children with GMFCS levels I to V because of its well-established psychometric properties and strong clinical utility.

   Pain for the adults CP Patients with intellectual and communicating disabilities will be assessed with the the Non-Communicating Adults Pain Checklist (NCAPC).
4. Parental interview.

In order to better define the subjects' pain status a parental interview will also be obtained. Parents are invited to report the presence, localization, etiology and duration of the subject's pain and to give information concerning the use of pain management measures. In children and adults without adequate communication parental experience will be recorded by a structured interview based on Paediatric Pain Profile (PPP) where the parent is invited a) to give a pain history and b) to answer questions in terms of non verbal learned reactions and behaviours to chronic pain on behalf of the subject (baseline assessments). The Paediatric Pain Profile is a tool that has been developed specially to help in assessing and monitoring pain in children with severe neurological impairments, especially those with impairments which lead them to be unable to communicate pain through speech. Such impairments mean that the children are dependant on their caregivers for interpretation of their signs of pain. It and has been used with adults up to 76 years of age. In order to better define the subjects' pain status we will take advantage of additional information from the young participants' medical record. In addition each case will be judged separately in terms of pain expression and severity, by a interdisciplinary panel of experts consisting of a general practitioner, a neurologist, a paediatrician, an orthopaedic, a psychologist, a dentist, a physical therapist, a speech therapist, an occupational therapist an expertise nurse, a social worker and the caregiver of the subject, who are daily involved in patient health needs and activities of living during their half day stay in the setting (Cerebral Palsy Greece) for at least 6 months. This group is going to consider for each patient the following questions:

1. What is the extent of the patient's disease or injury (physical impairment)?
2. What is the magnitude of the illness? That is, to what extent is the patient suffering, disabled, and unable to enjoy usual activities?
3. Does the individual's behaviour seem appropriate to the disease or injury, or is there any evidence of symptom amplification for any of a variety of psychological or social reasons (e.g. benefits such as positive attention, mood-altering medications, financial compensation)?

Aims of statistical analysis:

Agreement rates between different evaluation levels of chronic pain assessment will be examined permitting to determine the reliability level of various sources of information concerning the diagnosis of chronic pain in cerebral palsy. Further statistical analysis of check-list scores will attempt to identify items in these observational schedules that could be conceptualized as behavioural indicators of chronic pain in non-communicative subjects with cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

* Outpatients in the setting Cerebral Palsy Greece-Open Door. They all have a diagnosis of cerebral palsy.

Exclusion Criteria:

* All other subjects with or without a diagnosis of neurodevelopmental disorder.

Ages: 5 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Outpatients in Cerebral Palsy Greece-Open Door, an educational and therapeutic day care center in Athens for adults and children with cerebral palsy.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-16 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
Self-reported chronic pain (Intensity) -Children | Brief standardised procedure not exceding 5 minutes. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Score obtained by the administration of the Wong-Baker Faces Pain Rating Scale for children communicating participants .Minimum score:0 (no pain) Maximum score: 10 (pain of extreme intensity).
Self-reported chronic pain (Intensity)- Adults | Brief standardised procedure not exceding 5 minutes. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Score obtained by the administration of the Faces Pain Scale-Revised (FPS-R) for adult communicating participants. Minimum score:0 (no pain) Maximum score: 10 (pain of extreme intensity).
Self-reported chronic pain (location) | Βrief standardised procedure not exceding 5 minutes. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Location of self reported pain by communicating participants using the codification system of the Body Diagram
Chronic pain reported by caregiver (intensity) | Data obtained through questionnaire completed by caregiver at the participant's residence. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Score at pain intensity rating scale Minimum score 0: no pain Maximum score:10 (extreme pain)
Chronic pain in children non-communicating participants assessed by proxy (checklist) | 2 hour time frame required for completion of assessment procedure. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Total score obtained at the NCCPC- R (Non-Communicating Children's Pain Checklist). Minimum score:0 Maximum score: 90 Cut-off score is 7. A score higher than 7 signifies that the observed participant experiences chronic pain.
Chronic pain in adult non-communicating participants assessed by proxy (checklist) | 2 hour time frame required for completion of assessment procedure. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Total score obtained at the NCAPC (Non-communicating Adult Pain Checklist). Minimum score:0 Maximum score: 54 Cut- off score is 7. A score higher than 7 signifies that the observed participant experiences chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pantelis Stathis, MD PhD, Study Director — Cerebral Palsy Greece - Open Door
Locations (1):
- Cerebral Palsy Greece- Open Door, Athens, Greece